CLINICAL TRIAL: NCT02752633
Title: A Novel Assay for the Determination of Urinary 2,8-Dihydroxyadenine and Other Key Urinary Purine Metabolites: Effect of Allopurinol and Febuxostat on Urinary 2,8-Dihydroxyadenine Excretion in APRT Deficient Patients
Brief Title: Effect of Allopurinol and Febuxostat on Urinary 2,8-Dihydroxyadenine Excretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDCRN Protocol #6412; 2013-000975-33 (EudraCT Number); U54DK083908 (NIH)
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2017-12

CONDITIONS: Adenine Phosphoribosyltransferase Deficiency
Keywords: Xanthine dehydrogenase inhibitor treatment, pharmacotherapy
MeSH Terms: conditions — Adenine phosphoribosyltransferase deficiency | interventions — Allopurinol; Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study subjects (Experimental): Following a 7 day washout period all patients receive allopurinol (400 mg/day) as a single daily dose for 2 weeks. Following another 7 day washout period all participants receive febuxostat, 80 mg/day as a single daily dose, for 2 weeks.
  Interventions: Drug: Allopurinol; Drug: Febuxostat

INTERVENTIONS:
Drug: Allopurinol — This is a clinical trial comparing the effect of 80 mg/day of febuxostat to 400 mg/day of allopurinol on the urinary excretion of 2,8-dihydroxyadenine in patients with APRT deficiency.
  Other Names: Apurin; ATC Code M04AA01
Drug: Febuxostat — This is a clinical trial comparing the effect of 80 mg/day of febuxostat to 400 mg/day of allopurinol on the urinary excretion of 2,8-dihydroxyadenine in patients with APRT deficiency.
  Other Names: Uloric; ATC Code M04AA03

SUMMARY:
This exploratory pilot study was an open-label, crossover, single-center and non-randomized clinical trial designed to compare the effect of the standardly employed doses of allopurinol (400 mg/day) and febuxostat (80 mg/day) on the urinary 2,8-dihydroxyadenine (DHA) excretion in patients with adenine phosphoribosyltransferase (APRT) deficiency.

DETAILED DESCRIPTION:
This exploratory pilot study was an open-label, crossover, single-center and non-randomized clinical trial designed to compare the effect of the standardly employed doses of allopurinol (400 mg/day) and febuxostat (80 mg/day) on the urinary DHA excretion in patients with APRT deficiency. The study was conducted between May 2013 and May 2015 as participants were enrolled at different times. The only study site was Landspitali - The National University Hospital of Iceland in Reykjavik, Iceland. The Data (Observational) Safety Monitoring Board (D/OSMB) constituted by the National Institutes of Health had oversight responsibility of the Data Safety Monitoring Plan for this clinical trial. The monitoring board reviewed accrual, patterns and frequencies of all adverse events, and protocol compliance every 6-12 months. All study subjects gave a written informed consent for their participation.

Study participants were recruited from a group of patients with confirmed APRT deficiency enrolled in the National Institutes of Health supported APRT Deficiency Registry of the Rare Kidney Stone Consortium (RKSC, http://www.rarekidneystones.org/). Confirmation of APRT deficiency was based upon the determination of known biallelic pathogenic APRT mutations or absent APRT enzyme activity. Participants were eligible for inclusion if they a) were currently receiving allopurinol therapy (the currently recommended treatment for patients with APRT deficiency); b) were willing to interrupt their allopurinol treatment for a total of 3 weeks as outlined below and c) were at least 18 years of age. There were no other exclusion criteria if the above inclusions criteria were met.

Study interventions After a 7-day washout period, all consenting subjects were prescribed 400 mg of allopurinol in a single daily dose for 14 days. After a second 7-day washout period, all subjects were prescribed 80 mg febuxostat in a single daily dose for another 14 days. Twenty-four hour and first morning urine samples were collected at the end of the first washout period, and at the end of allopurinol and febuxostat treatment periods, respectively (days 7, 21 and 42). To minimize the potential adverse effect of dietary purine intake on the results, participants were asked to keep a food record while they collected the first 24 hr urine sample and adhere to the same diet when they collected the other two 24 hr urine samples. No further measures were taken to control dietary purine intake during the study period. At the end of the study, all patients were advised to return to their regular allopurinol dosing regimens.

Measurements Urinary DHA was measured using a rapid and robust ultra high power liquid chromatography - electrospray tandem mass spectrometry (UPLC-MS/MS)), recently developed by our group. The 24-hour urinary DHA excretion (mg/24-hours) was measured and the urinary DHA-to-creatinine ratio (mg/mmol) in first morning urine samples was calculated. Urine and serum creatinine concentrations were measured with an isotope dilution mass spectrometry (IDMS) standardized laboratory method.

Outcome measures The primary trial endpoint is the 24 hr urinary DHA excretion and in patients taking the two study drugs, allopurinol (daily dose 400 mg) and febuxostat (daily dose 80 mg), evaluated at the conclusion of each 14 day drug treatment period.

Statistical Analysis Data are presented as urinary DHA excretion (mg/day) for timed collections and urinary DHA-to-creatinine ratio in first morning urine samples. Data for the whole group are presented as a median (range). Differences in the median urinary DHA excretion and the urinary DHA-to-creatinine ratio, off pharmacotherapy and on the two study drugs, febuxostat and allopurinol, were compared with a paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 year and older who are enrolled in the APRT Deficiency Registry of The Rare Kidney Stone Consortium.

Exclusion Criteria:

* Patients do not want to interrupt drug (allopurinol) treatment for a total of two weeks as requested in protocol. No other exclusion criteria if inclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vidar O Edvardsson, MD, Principal Investigator — Landspitali - The National University Hospital of Iceland, Reykjavik
Locations (1):
- Landspitali - The National University Hospital of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Published in Eur J Intern Med. 2017 Dec 11, 2017. PMID: 29241594 DOI: 10.1016/j.ejim.2017.10.007
URL: http://www.sciencedirect.com/science/article/pii/S0953620517304156

REFERENCES:
- [Result] Runolfsdottir HL, Palsson R, Agustsdottir IM, Indridason OS, Edvardsson VO. Kidney Disease in Adenine Phosphoribosyltransferase Deficiency. Am J Kidney Dis. 2016 Mar;67(3):431-8. doi: 10.1053/j.ajkd.2015.10.023. Epub 2015 Dec 25. PMID 26724837
- See also: Official website of the Rare Kidney Stone Consortium — http://www.rarekidneystones.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Allopurinol/Febuxostat Treatment: This is a clinical trial comparing the effect of 80 mg/day of febuxostat to 400 mg/day of allopurinol on the urinary excretion of 2,8-dihydroxyadenine in patients with APRT deficiency.
Period: Overall Study
Arm/Group | Allopurinol/Febuxostat Treatment
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Allopurinol/Febuxostat Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 0
  Race: White | 9
  Race: More than one race | 0
  Race: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Iceland | 9

OUTCOME MEASURES:

1. Primary Outcome: Urinary 2,8-dihydroxyadenine Excretion
Time Frame: 7, 21 and 42 days
Measure: Median (Full Range); unit: mg/24-h
Groups:
- Allopurinol/Febuxostat Treatment: Following a 7 day washout period all patients receive allopurinol (400 mg/day) as a single daily dose for 2 weeks. Following another 7 day washout period all participants receive febuxostat, 80 mg/day as a single daily dose, for 2 weeks.
  Allopurinol: This is a clinical trial comparing the effect of 80 mg/day of febuxostat to 400 mg/day of allopurinol on the urinary excretion of 2,8-dihydroxyadenine in patients with APRT deficiency.
  Febuxostat: This is a clinical trial comparing the effect of 80 mg/day of febuxostat to 400 mg/day of allopurinol on the urinary excretion of 2,8-dihydroxyadenine in patients with APRT deficiency.
Arm/Group | Allopurinol/Febuxostat Treatment
Number analyzed (Participants) | 8
mg/24-h
  Baseline | 116 [75 to 289]
  On allopurinol treatment | 45 [13 to 112]
  On febuxostat treatment | 13 [10 to 13]
Statistical Analysis 1: Comparison: Allopurinol/Febuxostat Treatment; Data are presented as the urinary DHA excretion (mg/24 hr) and as the DHA-to-creatinine ratio (mg/mmol) in first morning void urine samples. Data are presented as a median (range). Differences in the median urinary DHA excretion and the urinary DHA-to-creatinine ratio between periods off pharmacotherapy and on the two study drugs, febuxostat and allopurinol, were assessed using the Wilcoxon signed rank test; Test type: Other; p < .05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Throughout the study, 42 days.
Arm/Group | Allopurinol/Febuxostat Treatment
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No